CLINICAL TRIAL: NCT02738957
Title: Effect of Prenatal Counseling on Breastfeeding Rates in Twins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria de Lourdes Brizot, Dr, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1131/09
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prenatal Counseling Group (Other): Patients in the PCG will receive specific counseling on breastfeeding consisting of three different counseling sessions during prenatal visits given by one two midwives involved in the study. The information will include: breastfeeding importance; how to prepare the nipples and breast for breastfeeding; the main complications and difficulties during the breastfeeding process and how to identify and overcome them; breastfeeding techniques and alternative positions for the simultaneous breastfeeding of twins, for example, "double cradle", "cradle-football" or "double-football", using illustrations and hands-on demonstration with doll models. During the counseling sessions patients will have the opportunity to discuss questions on breastfeeding.
  Interventions: Behavioral: Prenatal Counseling Group
- Control Group (No Intervention): No breastfeeding counseling during the antenatal period will be provided. The Control Group will receive non-specific counseling with standard orientation regarding breastfeeding after delivery and during their postpartum hospitalization period. This standard orientation will be provided by one of the midwives of the hospital during a single counseling session with brief guidance covering the following topics: starting breastfeeding, hygiene, infants' conditions, colostrum/breast milk, infants' positions, duration of breastfeeding, frequency of feeds, mammary milking, and stopping breastfeeding.

INTERVENTIONS:
Behavioral: Prenatal Counseling Group — Specific counseling on breastfeeding consisting of three different counseling sessions during prenatal visits given by one of the two midwives involved in the study. The information provided include the following: breastfeeding importance; how to prepare the nipples and breast for breastfeeding; the main complications and difficulties during the breastfeeding process and how to identify and overcome them; breastfeeding techniques and alternative positions for the simultaneous breastfeeding of twins, for example, "double cradle", "cradle-football" or "double-football", using illustrations and hands-on demonstration with doll models.
  Arms: Prenatal Counseling Group

SUMMARY:
Few studies have investigated breastfeeding in twins, and none have addressed the effect of antenatal counseling on breastfeeding twins.The purpose of this study is to investigate the effect of antenatal breastfeeding counseling on the breastfeeding rates in twin pregnancies.

DETAILED DESCRIPTION:
In singleton pregnancies, three randomized studies have recently examined the influence of antenatal breastfeeding education on the breastfeeding rates (Su et al. 2007; Mattar et al. 2007; Wong et al. 2014). Two of these studies did not find differences in the total breastfeeding rates between the groups that received and did not receive antenatal breastfeeding education at the infants' age of 6 months old (Su et al. 2007; Wong et al. 2014). However, Su et al. found higher exclusive breastfeeding rates for 6-months-old infants in the group that received antenatal counseling. In contrast, Mattar et al. 2007 found significantly difference in breastfeeding rates with individual counseling compared to non-counseling or only breastfeeding educational material with no counseling.

Few studies have investigated breastfeeding in twins specifically, and even fewer have focused on the duration of breastfeeding of twin infants. Furthermore, in our literature search, we did not find studies of breastfeeding of twins investigating the effect of antenatal education on breastfeeding twins. Our hypothesis is that mothers of twins receiving specific antenatal counseling on breastfeeding should have a higher rate of breastfeeding than mothers who do not receive antenatal breastfeeding counseling. Therefore, the purpose of this study was to investigate the effect of specific antenatal breastfeeding counseling on the breastfeeding rates in twin pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* twin pregnancies with both fetuses alive between 18 and 34 weeks of gestational age and followed at our twin clinic; absence of absolute contraindications for breastfeeding, such as positive serology for HIV, HTLV; absence of use of lactation inhibitors to treat prolactinoma, such as cabergoline and bromocriptine; and absence of major malformation of one or both twins that could preclude breastfeeding, including gastrointestinal defects, cleft lip and cleft palate, or malformations that would require neonatal surgery with prolonged hospital stay.

Exclusion Criteria:

* fetal or postnatal death of one or both twins; delivery before 32 weeks; major malformation diagnosed postnatal; and lost to follow up or no breastfeeding information.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Mother´s total and exclusive breastfeeding rates | 5 years
  Comparison of mothers' total and exclusive breastfeeding rates between the Prenatal Counseling Group (PCG) and Control Group (CG) in the three evaluated periods (30-40-days-old infants, 90-days-old infants and 180-days-old infants.

SECONDARY OUTCOMES:
Twin infant´s breastfeeding rates | 5 years
  Comparison of the rates of twin infant breastfeeding rates between the PCG and CG until 180 days of infants' age.For this analysis, the data of patients who were still breastfeeding at 180 days of infants' age will be censored at the time of the last obtained information.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA DE LOURDES BRIZOT, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No data will be shared

REFERENCES:
- [Background] Mattar CN, Chong YS, Chan YS, Chew A, Tan P, Chan YH, Rauff MH. Simple antenatal preparation to improve breastfeeding practice: a randomized controlled trial. Obstet Gynecol. 2007 Jan;109(1):73-80. doi: 10.1097/01.AOG.0000249613.15466.26. PMID 17197590
- [Background] Su LL, Chong YS, Chan YH, Chan YS, Fok D, Tun KT, Ng FS, Rauff M. Antenatal education and postnatal support strategies for improving rates of exclusive breast feeding: randomised controlled trial. BMJ. 2007 Sep 22;335(7620):596. doi: 10.1136/bmj.39279.656343.55. Epub 2007 Aug 1. PMID 17670909
- [Background] Wong KL, Tak Fong DY, Yin Lee IL, Chu S, Tarrant M. Antenatal education to increase exclusive breastfeeding: a randomized controlled trial. Obstet Gynecol. 2014 Nov;124(5):961-968. doi: 10.1097/AOG.0000000000000481. PMID 25437725
- [Derived] Mikami FC, de Lourdes Brizot M, Tase TH, Saccuman E, Vieira Francisco RP, Zugaib M. Effect of Prenatal Counseling on Breastfeeding Rates in Mothers of Twins. J Obstet Gynecol Neonatal Nurs. 2017 Mar-Apr;46(2):229-237. doi: 10.1016/j.jogn.2016.10.005. Epub 2017 Jan 5. PMID 28063805